CLINICAL TRIAL: NCT07169890
Title: Clinical Insights Into Dextrose Phonophoresis on Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005946
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dextrose Phonophoresis (Experimental): An individually prepared and equivalent 4-g dose of 0.33% dexamethasone gel (Vann Healthcare Services Inc, Glasgow, KY) from the same lot was applied. A topical dexamethasone gel applied then ultrasound treatment
  Interventions: Other: Dextrose Phonophoresis
- Ultrasound (Experimental): Using an ultrasound device set to a frequency of 1 MHz, with an intensity ranging from 0.5 to 1.5 W/cm², the ultrasound probe is moved in a circular motion over the skin for a duration of 5 to 10 minutes per session.
  Interventions: Other: Ultrasound
- Dextrose topical gel (Experimental): Topical application of dextrose gel
  Interventions: Other: Dextrose Topical application
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Dextrose Phonophoresis — To apply Dextrose Phonophoresis on a patient with acne vulgaris, begin by cleansing the affected skin area thoroughly with a gentle, non-comedogenic cleanser to remove any dirt or oils. Pat the skin dry with a clean towel. Prepare a dextrose gel, a 10% dextrose gel, which is then coupled with low-frequency ultrasound to facilitate deeper penetration of the dextrose
  Arms: Dextrose Phonophoresis
Other: Ultrasound — the ultrasound probe is moved in a circular motion over the skin for a duration of 5 to 10 minutes per session
  Arms: Ultrasound
Other: Dextrose Topical application — Apply a thin layer of the dextrose gel evenly across the acne-affected areas using a sterile applicator or cotton pad
  Arms: Dextrose topical gel

SUMMARY:
Acne vulgaris is a common cutaneous inflammatory disorder of the pilosebaceous unit, which runs a chronic course. The condition commonly manifests with papules, pustules, or nodules primarily on the face, although it can also affect the upper arms, trunk, and back. The pathogenesis of acne vulgaris involves the interaction of multiple factors that ultimately lead to the formation of its primary lesion, which is known as "comedo" (see Image. Acne Vulgaris). Although acne vulgaris is commonly observed among adolescents, it is not restricted to this age group and can affect individuals of various ages. The severity of this condition can vary, ranging from a mild presentation with only a few comedones to more severe forms characterized by disfiguring inflammatory manifestations, which can lead to hyperpigmentation, scarring, and adverse psychological effects.

DETAILED DESCRIPTION:
Dextrose phonophoresis emerges as a novel therapeutic modality in the management of mild to moderate acne vulgaris, an inflammatory skin condition that affects a significant portion of the adolescent and adult population. The rationale for employing dextrose phonophoresis lies in its dual mechanism of enhancing drug delivery and providing anti-inflammatory effects. Phonophoresis, which involves the use of ultrasound waves to enhance the transdermal delivery of topically applied medications, can potentiate the penetration of dextrose into the skin. Dextrose, a simple sugar, is hypothesized to modulate local inflammation and promote healing. This method leverages the mechanical effects of ultrasound to increase the permeability of the stratum corneum, thereby facilitating deeper penetration of dextrose into the dermal layers where it can exert its therapeutic effects.

The anti-inflammatory properties of dextrose are pivotal in its role in treating acne vulgaris. Acne is characterized by the inflammation of pilosebaceous units, and dextrose is believed to mitigate this inflammation through osmotic and possibly metabolic pathways. By reducing the inflammatory response, dextrose phonophoresis may decrease the erythema and lesion count associated with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 30 years.
* Clinically diagnosed with mild to moderate acne vulgaris.
* Willingness to comply with the study protocol and attend all treatment sessions.
* Medical Clearance: Participants must have medical clearance to participate in this study.

Exclusion Criteria:

* Individuals with severe acne vulgaris or other dermatological conditions affecting the face.
* Current use of systemic acne medications or topical treatments other than the study intervention.
* Known allergy to magnesium or ultrasound gel.
* Pregnant or breastfeeding individuals.
* Severe Comorbidities: Individuals with severe cardiovascular, pulmonary, metabolic, or vascular diseases
* Medication Interference: Individuals using medications known to affect presence of acne.
* Acute Psychological Conditions: Participants with acute psychological conditions that may interfere with participation or assessments.
* Obese patient whose BMI ≥ 30.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Acne Global Severity Scale (AGSS): | at baseline and at 4 weeks
  The Acne Global Severity Scale is a qualitative tool used to evaluate the overall severity of a patient's acne.Based on the examination, acne severity is classified into a standardized scale:((0: Clear skin with no inflammatory or non-inflammatory lesions,1: Almost clear with rare non-inflammatory lesions and no more than one small inflammatory lesion,2: Mild presence of non-inflammatory lesions with few inflammatory lesions,3: Moderate presence of numerous non-inflammatory lesions and several inflammatory lesions,4: Severe presence of many non-inflammatory and inflammatory lesions, including nodules).0-1: Represents mild or no acne; often considered within normal limits.2-4: Indicates increasing severity needing clinical intervention.
Acne Severity Index (ASI): | at baseline and at 4 weeks
  The Acne Severity Index is a quantitative measure that combines lesion counts and types to produce a single score.Score Calculation: Use the following formula to calculate the ASI :(( ASI = (Number of Comedones) + (2 × Number of Papules) + (3 × Number of Pustules) + (4 × Number of Nodules)).Scores can vary significantly; typically, lower scores (<10) indicate mild acne, while higher scores (20+) suggest moderate to severe acne.
Total Lesion Count (TLC) | at baseline and at 4 weeks
  Total Lesion Count is a straightforward quantitative assessment: Counting: Count all types of acne lesions (comedones, papules, pustules, nodules) on the face, chest, and back.(0-10 lesions: Considered mild,11-25 lesions: Moderate severity,26+ lesions: Severe acne requiring intervention).

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt